CLINICAL TRIAL: NCT04338711
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, PARTIAL CROSSOVER STUDY TO EVALUATE THE PHARMACOKINETICS AND SAFETY OF THREE AGE-APPROPRIATE MODIFIED RELEASE FORMULATIONS AND THE IMMEDIATE RELEASE SOLUTION OF TOFACITINIB IN HEALTHY ADULT VOLUNTEERS
Brief Title: A Study In Adult Healthy Volunteers To Asses Once Daily (QD) Dosing With The Selected Age-Appropriate Modified Release (MR) Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3921262
Record Dates: First submitted 2020-03-11; First posted 2020-04-08 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Single oral 10 mg dose of tofacitinib MR E1 administered in the fasted state.
  Interventions: Drug: tofacitinib modified release (MR)
- Treatment B (Experimental): Single oral 10 mg dose of tofacitinib MR E2 administered in the fasted state.
  Interventions: Drug: tofacitinib modified release (MR)
- Treatment C (Experimental): Single oral 10 mg dose of tofacitinib MR E3 administered in the fasted state.
  Interventions: Drug: tofacitinib modified release (MR)
- Treatment D (Experimental): Single oral 10 mg dose of tofacitinib MR E1 administered in the fed state.
  Interventions: Drug: tofacitinib modified release (MR)
- Treatment E (Experimental): Single oral 10 mg dose of tofacitinib MR E3 administered in the fed state.
  Interventions: Drug: tofacitinib modified release (MR)
- Treatment F (Active Comparator): Single oral 10 mg dose of tofacitinib IR Solution (10 mL of the 1 mg/mL solution) administered in the fasted state.
  Interventions: Drug: tofacitinib modified release (MR)

INTERVENTIONS:
Drug: tofacitinib modified release (MR) — Single oral 10 mg multi particulate dose of dose of tofacitinib MR with different levels of enteric coating (MR E1, MR E2, and MR E3) in the fasted state. Additionally, the lowest and highest enteric coating levels will also be evaluated in the fed state.
  Treatment F: a 10 mg oral dose of tofacitinib IR solution

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) and safety of an age-appropriate tofacitinib Modified Release (MR) formulation with varying level of enteric coating. The effect of food on the PK of age-appropriate tofacitinib MR formulation with the lowest and higher levels of enteric coating will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

  1. . Achieved postmenopausal status, defined as: cessation of regular menses for at lease 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
  2. . have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. . have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight ˃50 kg (110 lbs) for males and ˃45 kg (99 lbs) for females
* No evidence of active or latent or inadequately treated infection with Mycobaceterium tuberculosis (TB)

Exclusion Criteria:

* Evidence or history of clinical significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, season allergies at the time of dosing.
* Clinically significant infections within the past 3 months (for example, those requiring hospitalization or parenteral antibiotics, or as judged by the investigator), evidence of any infection within the past 7 days, history of disseminated herpes simplex infection or recurrent (˃1 episode) herpes zoster or disseminated herpes zoster.
* Absolute lymphocyte count at Screening or Baseline (Day -1 of Period 1) less than the lower limit of the reference range for the local laboratory (lymphocyte count ˂0.8* 10˄3).
* Evidence of hematopoietic disorder or hemoglobin ˂12.5 g/dL for females and ˂13 g/dL for males at Screening or Baseline ((Day -1 of Period 1).
* Evidence or history of cyclic neutropenia.
* Personal or family history of hereditary immunodeficiency (eg, severe combined immunodeficiency disorder [SCID], Wiskott-Aldrich syndrome, X-linked agammaglobulinemia).
* Vaccination with live or attenuated vaccines within 6 weeks of dosing, or is to be vaccinated with these vaccines at any time during study treatment or within 6 weeks following discontinuation of dosing.
* Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
* History of, or current positive results for any of the following serological tests: human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatits B surface antigen (HepBsAg), Hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
* Malignancy or a history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Positive urine drug test.
* History of regular alcohol consumption.
* Use of tobacco-or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of the investigational product (whichever is longer).
* Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval ˃450 msec or a QRS interval ˃120 msec.
* Nursing females or females of childbering potential. Male subjects who are unwilling or unable to use a condom plus a highly effective method of contraception as outline in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of investigational product.
* Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or inducers (eg, phenytoin, carbamazepine, rifampin) within 14 days or 5 half-lives (whichever is longer) prior to dosing.
* Consumption of grapefruit or grapefruit-related citrus fruits (eg, Seville oranges, pomelos) or juices within 7 days prior to dosing.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparing-induced thrombocytopenia.
* History of hypersensitivity to tofacitinib or any of the components of the formulation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] (AUCinf ) | 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of Modified Release (MR) formulation compared to Immediate Release (IR) solution
Maximum Observed Plasma Concentration (Cmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Maximum (or peak) plasma concentration of MR formulation compared to IR solution
Time to Reach Maximum Observed Plasma Concentration (Tmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Maximum time to peak plasma concentration of MR formulation compared to IR solution

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Through study completion, approximately 3 months
  The incidence of all-causality TEAEs is summarized by System Organ Class (SOC) and MedDRA preferred term
  Treatment-Emergent Adverse Events (Treatment Related)
  For each AE, the investigator will pursue and obtain information adequate both to determine the outcome of the AE and to assess whether it met the criteria for classification as a serious adverse event (SAE)
Number of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Leading to Discontinuation | Through study completion, approximately 3 months
  Discontinuations from the study or study treatment due to AEs, temporary discontinuations or dose reductions due to AEs reported during the study
Number of Participants With Clinically Significan Change from Baseline in Physical Examination Findings | Through study completion, approximately 3 months
  Full Physical examination includes examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. A limited or abbreviated physical examination assesses the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings are considered to be clinically significant based on investigator's assesment.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Through study completion, approximately 3 months
  The following parameters will be analyzed for examination of vital signs: oral temperature, supine blood pressure, pulse rate.
Number of Participants with Clinically Significant Change in the QTC interval from Baseline in 12-lead ECGs | Through study completion, approximately 3 months
  Criteria for potential clinical concern in ECG parameters: maximum corrected QT interval (QTc) from baseline is greater than or equal in range of 45 millisecond (msec); or an absolute QTc value of greater than or equal in range of 500 msec in any scheduled ECG.
Number of Participants with Clinically Significant Laboratory Abnormalities | Through study completion, approximately 3 months
  The following parameters will be analyzed for laboratory examination: hematology, chemistry, urinalysis, microsopy [only if urine dipstick is positive for blood, protein, nitrites or leukocyte esterase]; other [only at screening] serum follicle stimulating hormone ) for female subjects only who are amenorrheic for at least 12 consecutive months), urine drug testing hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, HIV, QuantiFERON Gold test. Clinical significance of laboratory parameters will be determined at the investigator's discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921262